CLINICAL TRIAL: NCT03564860
Title: His Bundle Pacing Device Electrogram Data Collection
Brief Title: HBP Device EGM Data Collection
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10234
Record Dates: First submitted 2018-05-15; First posted 2018-06-21 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Sick Sinus Syndrome; AV Block; Heart Failure
MeSH Terms: conditions — Sick Sinus Syndrome; Atrioventricular Block; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HBP device data collection group: Device electrograms and 12-lead ECG will be collected from patients over the age of 18 years who have been previously implanted with a permanent His Bundle pacing lead and an Abbott pacemaker, defibrillator, or cardiac resynchronization therapy device during a standard-of-care device follow-up visit.
  Interventions: Procedure: Device data collection

INTERVENTIONS:
Procedure: Device data collection — Collection of device electrograms and 12-lead ECG during a device follow-up visit

SUMMARY:
This is a single-arm, non-randomized, non-blinded study designed to collect device data in patients with permanent His bundle (HB) pacing lead and an existing Abbott permanent pacemaker, defibrillator, or cardiac resynchronization device. Prospective data collection includes surface electrocardiograms, intracardiac electrograms, and pacing parameters, recorded during a patient visit. Additional retrospective data collection includes procedural data during the HB pacing lead and device implant.

Up to 200 subjects will participate in this clinical investigation. The clinical investigation will be conducted at up to 8 centers worldwide.

The total duration of the clinical investigation is expected to be 1 year, including enrollment and data collection from all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Has previously implanted with Abbott device and any pacing lead at HB
* Age ≥ 18 years
* Ability to provide informed consent for study participation
* Willing to comply with study evaluation requirements

Exclusion Criteria:

* Suspected pacing system failure
* Lead impedance out of range
* Ventricular sensing amplitude lower than 0.5 mV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intended population for this clinical investigation consists of patients over the age of 18 years who have been previously implanted with a permanent His Bundle pacing lead and an Abbott pacemaker, defibrillator, or cardiac resynchronization therapy device.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Amplitude of device electrogram | through study completion, an average of 1 year
  Mean amplitude of device electrogram during His bundle pacing
Duration of device electrogram | through study completion, an average of 1 year
  Mean duration of device electrogram during His bundle pacing

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - *Heart Center Research, LLC., Huntsville, Alabama
  - Donald Guthrie Foundation for Education & Research, Sayre, Pennsylvania
  - Greenville Health System, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No